CLINICAL TRIAL: NCT01694342
Title: Telomere Parameters Like Telomere Length, Telomerase Expression, Telomere Capture and Aneuploidy in Patients With Nonalcoholic Fatty Liver
Brief Title: Telomere Parameters in Patients With Nonalcoholic Fatty Liver
Acronym: telomereFL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ramona 1.0
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-07

CONDITIONS: FATTY LIVER; NO MALIGNANCY; NO DECOMPENSATED ILLNESS
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Telomerase, through its regulatory function on telomere length may play an important role in immune function, cellular replicative life span, and carcinogenesis. Non-alcoholic fatty liver disease (NAFLD) is considered a benign condition, but in some cases, it may progress to cirrhosis and hepatocellular carcinoma. The risk factors for that evolution are not fully understood.

Our group showed in a previous study, that hTERT mRNA expression is lower in peripheral lymphocytes of patients with fatty liver, compared to healthy controls. This finding could explain the telomere shortening found previously in these patients by our group [20] and others [21]. Furthermore, we found higher rates of TC in these patients, probably due to an attempt to counteract the shortening of the telomeres and to stabilize them. This is through a different mechanism that is not telomerase-mediated.

Telomere capture is considered an alternative way to maintain telomere length and chromosomal stability [3]. It is a more common mechanism for chromosome stabilization and repair, in contrast to the telomerase-mediated process of chromosome healing and elongation This study aimed to evaluate mechanisms of telomere homeostasis like telomere shortening, telomerase activity, telomere capture and aneuploidy in patients with NAFLD in order to explain previous findings of telomere shortening in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* diagnosis of fatty liver

Exclusion Criteria:

* no malignancy
* no eligible to sign the consent paper

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals - over 18 years old that were diagnosed with nonalcoholic fatty liver and are on follow-up in our liver unit
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-09

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Hospital, Kfar Saba, Israel